CLINICAL TRIAL: NCT03509883
Title: A Study to Assess the Absorption of Apixaban (BMS-562247) Sprinkle Capsules Compared With Tablets in Healthy Volunteers
Brief Title: Bioavailability of Apixaban Sprinkle Compared to Apixaban Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV185-687
Record Dates: First submitted 2018-04-18; First posted 2018-04-26 (Actual); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apixaban sprinkle capsules followed by apixaban tablets (Experimental): Apixaban (BMS-562247) sprinkle capsules followed by apixaban tablets
  Interventions: Drug: Drug: Apixaban sprinkle capsules; Drug: Experimental: Apixaban tablets followed by apixaban sprinkle capsules
- Apixaban tablets followed by apixaban sprinkle capsules (Active Comparator): Apixaban (BMS-562247) tablets followed by apixaban sprinkle capsules
  Interventions: Drug: Drug: Apixaban sprinkle capsules; Drug: Experimental: Apixaban tablets followed by apixaban sprinkle capsules

INTERVENTIONS:
Drug: Drug: Apixaban sprinkle capsules — Single dose (25 x 0.1 mg capsules), oral administration
  Other Names: •BMS-562247; •Eliquis
Drug: Experimental: Apixaban tablets followed by apixaban sprinkle capsules — Apixaban sprinkle capsules Single dose (25 x 0.1 mg capsules), oral administration
  Other Names: •BMS-562247

SUMMARY:
The purpose of this study is to evaluate the absorption of apixaban (BMS-562247) into the bloodstream of healthy volunteers, when administered as sprinkle capsules compared to tablets. Eligible participants will be randomly assigned to 1 of 2 treatment sequences and will receive a single oral dose of apixaban twice during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Healthy male and female participants determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead ECGs (electrocardiograms), vital signs and clinical laboratory determinations.
* Women of childbearing potential (WOCBP) must have negative serum pregnancy tests (performed at screening and Day 1), must not be breastfeeding, and must agree to follow instructions for method(s) of contraception for duration of treatment with study drug apixaban, and for a total of 33 days after last dose of apixaban.
* Males sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for duration of treatment with study drug apixaban, and for a total of 93 days after the last dose of apixaban; and must be willing to refrain from sperm donation during this time.
* Body mass index (BMI) of 18.0 to 30.0 kg/m², inclusive. Body mass index = weight (kg)/[height(m)]².

Exclusion Criteria:

* History of chronic headaches (occurring 15 days or more a month) over the previous 3 months.
* History of gastroesophageal reflux disease, dyspepsia, protracted nausea, or chronic diarrhea.
* History or evidence of abnormal bleeding or coagulation disorders, hypermenorrhea, intracranial hemorrhage, or abnormal bleeding or coagulation disorders.
* Inability to comply with restrictions and prohibited treatments (e.g. women currently taking hormonal contraception).
* Use of tobacco- or nicotine-containing products (e.g. cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, nicotine gum) within 6 months prior to study drug administration.
* Donation of blood to a blood bank or in a clinical study (except screening or follow-up visit) within 4 weeks of study drug administration (within 2 weeks for plasma only).

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 94 Participants Enrolled; 30 participants Randomized; Reasons Not Randomized: 43 participants no longer meet study criteria; 12 were lost to follow up 9 other; 5 screening extras: 4 back ups
Groups:
- Treatment A, Then Treatment B: Apixaban tablets (treatment A) followed by apixaban sprinkle capsules (treatment B)
- Treatment B, Then Treatment A: Apixaban sprinkle capsules (treatment B) followed by apixaban tablets (treatment A)
Period: Initial Treatment
Arm/Group | Treatment A, Then Treatment B | Treatment B, Then Treatment A
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Initial Treatment Washout
Arm/Group | Treatment A, Then Treatment B | Treatment B, Then Treatment A
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Cross-over and Treatment
Arm/Group | Treatment A, Then Treatment B | Treatment B, Then Treatment A
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment A: Apixaban tablets (treatment A) followed by apixaban sprinkle capsules (treatment B)
- Treatment B: Apixaban sprinkle capsules (treatment B) followed by apixaban tablets (treatment A)
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (7.6) | 32.8 (7.3) | 32.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentration as Measured by Maximum Observed Plasma Concentration (Cmax)
Description: Assessment of bioavailability of apixaban 0.5mg tablets relative to apixaban 0.1mg Sprinkle in terms of concentration
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: Apixaban tablets (treatment A)
- Treatment B: Apixaban sprinkle capsules (treatment B)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
ng/mL | 77.4 (26.5) | 99.3 (24.6)

2. Primary Outcome: AUC (0-T) - Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration
Description: Assessment of bioavailability of apixaban 0.5mg tablets relative to apixaban 0.1mg Sprinkle in terms of plasma concentration and time
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
ng*h/mL | 695.9 (27.3) | 769.2 (23.7)

3. Primary Outcome: AUC (INF) - Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time
Description: as for outcome 2
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
ng*h/mL | 714.7 (26.9) | 787.9 (23.1)

4. Secondary Outcome: Tmax - Time of Maximum Observed Plasma Concentration
Description: Assessment of bioavailability of apixaban 0.5mg tablets relative to apixaban 0.1mg Sprinkle in terms time of maximum concentration
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h (hours)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
h (hours) | 2.30 (36.4) | 0.98 (43.8)

5. Secondary Outcome: T-Half - Terminal Plasma Half Life.
Description: Assessment of bioavailability of apixaban 0.5mg tablets relative to apixaban 0.1mg Sprinkle in terms of time required to reach to half of plasma concentration
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h (hours)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
h (hours) | 8.81 (39.2) | 7.91 (32.7)

6. Secondary Outcome: Frel - Relative Bioavailability
Description: The relative bioavailability of 0.1mg apixaban sprinkle capsules as compared to 0.5mg tablet formulation
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Groups:
- Treatment B: Sprinkle Capsules as compared to tablet formulation
Arm/Group | Treatment B
Number analyzed (Participants) | 30
Percentage | 110.24 (9.3)

7. Secondary Outcome: Number of Participants With Adverse Events Regardless of Causality, Serious Adverse Events and Adverse Events Leading to Discontinuation
Description: Adverse events regardless of causality, Serious Adverse Events & Adverse events leading to discontinuation
Time Frame: Day 1 to Day 38
Population: All Treated Participants
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
Participants
  Adverse Events | 7 | 3
  Serious Adverse Events | 0 | 0
  Adverse Events leading to Discontinuation | 0 | 0

8. Secondary Outcome: Physical Measurement - Height
Description: Average height of all participants treated
Time Frame: Pre-treatment Screening
Population: All treated participants
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
centimeter (cm) | 173.23 (5.81) | 165.86 (8.86)

9. Secondary Outcome: Physical Measurement - Weight
Description: Average weight of all participants treated
Time Frame: Pre-treatment screening to Day 8
Population: All treated participants
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
kilograms (kg)
  Pre-treatment | 78.09 (5.81) | 165.86 (8.86)
  Day 1 | 77.83 (3.35) | 71.47 (12.55)
  Day 8 | 76.15 (11.60) | 70.64 (12.28)

10. Secondary Outcome: Physical Measurement - Body Mass Index (BMI)
Description: Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive. Body mass index = weight (kg)/[height(m)]2.
Time Frame: Pre-treatment Screening to Day 8
Population: All treated participants
Measure: Mean (Standard Deviation); unit: kilograms / Meters² (kg/m²)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
kilograms / Meters² (kg/m²)
  Pre-treatment | 22.96 (3.35) | 25.85 (2.91)
  Day 1 | 25.87 (3.50) | 25.84 (2.87)
  Day 8 | 25.31 (3.25) | 25.55 (2.79)

11. Secondary Outcome: Number of Participants With a Given Clinical Laboratory Abnormality
Description: Assessment of clinical laboratory abnormalities
Time Frame: Day 1 to Day 8
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
participants
  hemoglobin abnormal low | 0 | 0
  Hematocrit abnormal low | 0 | 0
  Platelet count abnormal low | 0 | 0
  platelet count abnormal high | 0 | 0
  Leukocytes abnormal low | 0 | 0
  Leukocytes Abnormal high | 0 | 0
  Neutrophils (Absolute) Abnormal low | 2 | 1
  Lymphocytes abnormal low | 0 | 0
  Lymphocytes Abnormal high | 0 | 0
  Monocytes (Absolute) Abnormal High | 0 | 0
  Basophils (absolute) Abnormal High | 0 | 0
  Eosinophils (absolute) Abnormal High | 0 | 0
  Prothrombin Time (PT) Abnormal High | 0 | 0
  International Normalized Ratio (INR) Abnormal High | 0 | 0
  Alkaline Phosphate (ALP) Abnormal High | 0 | 0
  Aspartate Aminotransferase (AST) Abnormal High | 0 | 0
  Alanine Aminotransferase (ALT) Abnormal High | 0 | 0
  Bilirubin, Total Abnormal High | 0 | 0
  Blood Urea Nitrogen (BUN) Abnormal High | 0 | 0
  Creatinine Abnormal High | 0 | 0
  Sodium Abnormal Low | 0 | 0
  Sodium, Serum Abnormal High | 0 | 0
  Potassium Abnormal Low | 0 | 0
  Potassium, Serum Abnormal High | 0 | 0
  Chloride, Serum Abnormal Low | 0 | 0
  Chloride, Serum Abnormal High | 0 | 0
  Calcium, Serum Abnormal Low | 0 | 0
  Calcium, Serum Abnormal High | 0 | 0
  Phosphorus, Inorganic Abnormal Low | 0 | 0
  Phosphorus, Inorganic Abnormal High | 0 | 0
  Glucose, Fasting Serum Abnormal Low | 0 | 0
  Glucose, Fasting Serum Abnormal High | 0 | 0
  Protein, Total Abnormal Low | 0 | 0
  Protein, Total Abnormal High | 0 | 0
  Albumin Abnormal Low | 0 | 0
  Lactate Dehydrogenase (LDH) Abnormal High | 0 | 0
  Protein, Urine Abnormal High | 0 | 0
  Glucose, Urine Abnormal High | 0 | 0
  Blood, Urine Abnormal High | 2 | 2
  WBC, Urine Abnormal High: number analyzed (Participants) | 6 | 5
  WBC, Urine Abnormal High | 2 | 2
  RBC, Urine Abnormal High: number analyzed (Participants) | 6 | 5
  RBC, Urine Abnormal High | 1 | 0

12. Secondary Outcome: Number of Participants With Out-of Range Vital Signs: Blood Pressure
Description: Number of participants with Out-of Range Blood Pressure changes as follows:
  Systolic Blood Pressure (SBP) mmHg < 90 and change from baseline < -20 > 140 and change from baseline > 20
  Diastolic Blood Pressure (DBP) mmHg < 55 and change from baseline < -10 > 90 and change from baseline > 10
Time Frame: Day 1 to Day 8
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
participants
  SBP < 90 and change from baseline < -20 | 0 | 0
  SBP >140 and change from baseline >20 | 0 | 0
  DBP < 55 and change from baseline < -10 | 0 | 1
  DBP >90 and change from baseline >10 | 0 | 0

13. Secondary Outcome: Number of Participants With Out-of Range Vital Signs: Heart Rate (Bpm)
Description: Number of participants with Out-of Range Heart Rate changes as follows:
  < 55 and change from baseline < -16 >100 and change from baseline > 10
Time Frame: Day 1 to Day 8
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
participants
  <55 and change from baseline < -16 | 0 | 0
  >100 and change from baseline > 10 | 0 | 0

14. Secondary Outcome: Number of Participants With Out-of Range Vital Signs: Respiration Rate
Description: Number of participants with Out-of Range respiration rate changes as follows:
  Respiration Rate is measured by number of respiration per min (rpm) > 16 rpm Change from baseline >10 rpm > 16 rpm or change from baseline > 10 rpm
Time Frame: Day 1 to Day 8
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
participants
  >16 rpm | 1 | 1
  change from baseline > 10 rpm | 0 | 0
  >16 or change from baseline >10 rpm | 1 | 1

15. Secondary Outcome: Number of Participants With Out-of Range Vital Signs: Temperature
Description: Number of participants with Out-of Range temperature changes as follows:
  Temperature is measured in Degrees centigrade (°C)
  >38.3°C Change from baseline > 1.6°C >38.3°C or change from baseline > 1.6°C
Time Frame: Day 1 to Day 8
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
participants
  >38.3°C | 0 | 0
  change from baseline > 1.6°C | 0 | 0
  >38.3°C or change from baseline > 1.6°C | 0 | 0

16. Secondary Outcome: Number of Participants With Out-of Range ECG Evaluations
Description: Number of participants with out-of-range ECG changes. ECG intervals are measured in milliseconds (msec)
Time Frame: Day 1 to Day 8
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
participants
  PR Interval Baseline ≤ 200 | 30 | 30
  PR Interval Baseline >200 | 0 | 0
  PR Interval Maximum on Treatment ≤ 200 | 29 | 30
  PR Interval Maximum on Treatment >200 | 1 | 0
  QRS Interval Baseline ≤ 120 | 30 | 30
  QRS Interval Baseline >200 | 0 | 0
  QRS Interval Maximum on Treatment ≤ 120 | 30 | 30
  QRS Interval Maximum on Treatment > 120 | 0 | 0
  QT Interval Baseline ≤ 500 | 30 | 30
  QT Interval Baseline >500 | 0 | 0
  QT Interval Maximum on Treatment ≤ 500 | 30 | 30
  QT Interval Maximum on Treatment > 500 | 0 | 0
  QT Interval Increase from Baseline ≤ 30 | 29 | 29
  QT Interval Increase from Baseline > 30 | 1 | 1
  QTcF Interval Baseline ≤ 450 | 30 | 30
  QTcF Interval Baseline >450 | 0 | 0
  QTcF Interval Maximum on Treatment ≤ 450 | 30 | 30
  QTcF Interval Maximum on Treatment > 450 | 0 | 0
  QTcF Interval Increase from Baseline ≤ 30 | 30 | 30
  QTcF Interval Increase from Baseline > 30 | 0 | 0

ADVERSE EVENTS:
Time Frame: 40 days (1st dose to 30 days after study completion)
Groups:
- Treatment A: Apixaban tablets 5 × 0.5-mg
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=30) | Treatment B (N=30)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03509883/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03509883/SAP_001.pdf